CLINICAL TRIAL: NCT06002282
Title: HPV Vaccine Confident Families
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: NIH grant termination
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Racquel Kohler, PhD, MSPH, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Pro2022001385; K22CA258675 (NIH); 132211 (Other: Rutgers, Cancer Institute of New Jersey)
Record Dates: First submitted 2023-07-31; First posted 2023-08-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Human Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tailored Messaging (Experimental): Tailored messages based on parents' HPV vaccine hesitancy and perceived barriers to vaccination.
  Interventions: Behavioral: Tailored messages
- Standard Messaging (Active Comparator): Standard (untailored) messages about HPV vaccination reminder/recall.
  Interventions: Behavioral: Standard messages

INTERVENTIONS:
Behavioral: Tailored messages — Messages will be individually tailored to parents' responses to a baseline survey (child gender, vaccination status) and real-time responses to interactive prompts about vaccine hesitancy determinants with links to additional information (e.g., CDC, NJ Department of Health) and community resources to overcome barriers.
  Arms: Tailored Messaging
Behavioral: Standard messages — Generic reminder/recall HPV vaccination messages.
  Arms: Standard Messaging

SUMMARY:
The objectives of the study are to pilot test a tailored intervention among Black families with adolescents. The hypotheses are that the study protocol will be feasible and messages tailored to parents' needs will increase vaccine confidence and intention to vaccinate.

ELIGIBILITY:
Inclusion Criteria:

* parent or legal guardian of at least one child aged 9-13 years who has received 0 or 1 dose of HPV vaccine;
* identify as Black or African American adult;
* have access to personal mobile phone and agree to send/receive MMS messages;
* able to speak and understand English; and
* able to provide informed consent to participate

Exclusion Criteria:

* parent or legal guardian of child outside of participation age range or who has completed multiple doses of HPV vaccine;
* does not identify as Black or African American adult;
* does not have personal mobile phone;
* unable to speak and understand English;
* not willing to consent to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment | After enrollment completion, 6 months
  ratio of parents recruited to potential parents approached to participate in study
Feasibility - Retention | Post intervention completion, 1 year
  ratio of parents completing post-intervention surveys to the number enrolled
Feasibility - Intervention Delivery | Two weeks after intervention begins
  ratio of parents receiving HPV message to the number enrolled
Feasibility - Intervention response | Two weeks after intervention completion
  assessment of how often participants completed hesitancy questions across the intervention period
Feasibility - Intervention utility | Two weeks after intervention completion
  Perceived ease of use, likeability, helpfulness, impact - Mobile App Rating Scale (1-inadequate, 2-poor, 3-acceptable, 4-good, and 5-excellent)

SECONDARY OUTCOMES:
Vaccine Intention | Immediately post-intervention (6 months)
  Parent reported intention to vaccinate adolescent in next 6 months
Vaccine Confidence | Immediately post-intervention (6 months)
  Parent-reported response to scale assessing benefits of vaccination, harms of vaccination, and trust in health care providers (1 - strongly disagree to 5 - strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Racquel Kohler, PhD, Principal Investigator — Rutgers
Locations (1):
- Rutgers, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No